CLINICAL TRIAL: NCT06147999
Title: Impact of a Biophoton Therapy on Patients With Brain Disorders
Acronym: Alzheimer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Institute of All Medicines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIAM-BD369
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Brain Disorders - Alzheimer's Disease, Dementia, Parkinson's Disease, Traumatic Brain Injury
Keywords: Alzheimer's Disease, and/or; dementia, and/or; Parkinson's Disease, and/or; Traumatic Brain Injury, and/or
MeSH Terms: conditions — Dementia; Parkinson Disease; Brain Injuries, Traumatic; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This study is a randomized, triple-blinded, placebo-controlled prospective intervention clinical research in two groups. About 80 patients with brain disorder will participate in the clinical interventional study at the hotel-like Tesla MedBed Center in Butler, PA, USA.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The 14 inactive Biophoton Generators packed with the same 32-Oz metal can as the active Treatment device will be labeled with a code and placed under a hotel bed for use. The shape, weight and overall looking is identical between the active and placebo devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment Group (Experimental): The 14 active Biophoton Generators packed with the same 32-Oz metal can will be labeled with a code and placed under a hotel bed. Each participant will rest on the bed during the entire study period for 4 weeks. Participants will receive biophotons inside of the biophoton field generated by 14 active Biophoton Generators
  Interventions: Device: Biophotonizer - a Biophoton Generator
- Control Group (Placebo Comparator): The 14 inactive Biophoton Generators packed with the same 32-Oz metal can will be labeled with a code and placed under a hotel bed. Each participant will rest on the bed during the entire study period for the first 2 weeks. Then will be switched to the active treatment group for being treated for 4 weeks. Participants will receive placebo effect from the 14 inactive comparators.
  Interventions: Device: Biophotonizer - a Biophoton Generator

INTERVENTIONS:
Device: Biophotonizer - a Biophoton Generator — A biophotonizer is a device producing strong biophoton field. These biophotons help the human body to gain self-healing capacity to heal many disorders, including brain disorders.

SUMMARY:
Previous clinical studies revealed that the newly developed biophoton therapy has been safe and effective in treating patients with Alzheimer's disease, dementia, stroke, traumatic brain injury, or Parkinson's disease. The current study is to confirm the previous clinical observation by conducting as a randomized, triple-blinded, placebo-controlled prospective intervention clinical research. About 80 patients with brain disorder (Alzheimer's disease, dementia, stroke, traumatic brain injury, Parkinson's disease) will participate in the intervention clinical study at the Tesla MedBed Center located in Butler, PA.

DETAILED DESCRIPTION:
The participant will live in the hotel-like research center for 4 weeks, or 6 weeks if the participants are randomly placed in a placebo group. The initial 2 weeks of participation is triple blinded to record the placebo effects, as each set of the study device is labelled with a unique code for use by only one participant. The change of the placebo device to the treatment device will be performed by the study device management team staff who will not inform the study participant nor study research staff who involve study data collection. Each participant assigned to the Control Group will be treated with 14 placebo devices under the bed plus two placebo devices to place in bed on each side of the head. Each participant assigned to the Treatment Group will receive 14 Biophoton generator devices under the bed plus two Biophoton Generators to place in bed on each side of the head. Each participant will use the Treatment or Control device for at least 8 hours every night for the first 2 weeks during sleep. During the day, participants are welcome to move around the facility, visit people or places. At the end of the first 2 weeks, the study participants will be advised whether she/he will be continually in a treatment group for 2 more weeks or be switched from a placebo group to a treatment group for 4 more weeks. Each participant will be guided by study team staff on their assigned testing day to answer the standard SF-36 questionnaires (SF-36) for measuring life quality, Cognitive Improvement Questionnaires, physician performed neurologic examination, Bio-well energy test, the Electroencephalography (EEG) test, blood flow test, and brain biophoton test, respectively at the baseline, 2 and 4 weeks after the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must meet conditions for approval.
* Must be 18-years or older and stay in a hotel.
* Must have a caregiver willing to support the participant's full involvement in the study. • The caregiver can assist in completing all study surveys.
* Can provide informed consent or can be assisted by caregiver.
* Can provide a clinical diagnosis of a brain disorder.
* Can complete all study procedures during the study.
* Must be fluent in English (or the Caregiver can fully translate).
* Women of childbearing age must provide results of a pregnancy test in order to participate.

Exclusion Criteria:

* Any untreated mental illnesses, that would affect study participation. This will be judged by the caregiver, or by the clinical study medical expert.
* Someone that relies on a ventilator.
* Someone who has a deep brain stimulator, pacemaker, or any implanted electronic devices.
* Co-morbid conditions that would interfere with study activities or response to treatment, which may include severe chronic pulmonary disease, history of uncontrolled seizures, acute or chronic infectious illness, severe diabetes, kidney failure, or any end-of-life prognosis.
* Is participating in another investigational drug or device trial.
* Has an active infectious disease, such as COVID-19.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-11-08 (Estimated); Study Completion 2026-11-08 (Estimated)

PRIMARY OUTCOMES:
Overall Life Quality impacted by Biophoton Therapy | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Short Form Health Survey (SF-36) will be used to assess life quality: scored from 0 (worst health) to 100 (best heath).
Cognitive Capacity impacted by Biophoton Therapy | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Montreal Cognitive Assessment (MOCA), Score below 10, severe cognition damage; 26-30, normal cognition.

SECONDARY OUTCOMES:
Neurological Examination impacted by Biophoton Therapy | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Neurological Examination by a Study Physician. The higher the score, the healthier the participant.
Brain function change impacted by Biophoton Therapy | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Brain function change is to be detected by using an EEG machine. Eye reaction time - the shorter the healthier.
Brain Bio-Energy impacted by Biophoton Therapy | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Using Bio-Well GDV Camera device and calculated by multiplication of areas of the brain. The more balanced joules, the better brain energy.
Blood Circulation impacted by Biophoton Therapy | 0-2 weeks, 0-4 weeks after starting the study treatment.
  FALCON QUAD measures circulation using the ankle-brachial index. The more balanced measurement, the better blood circulation.

OTHER OUTCOMES:
Safety of the Study participant impacted by Biophoton Therapy | 0-2 weeks, 0-4 weeks after starting the study treatment.
  Number of participants with treatment-related adverse events as assessed by CTCAEv4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tesla MedBed Center, 139 Pittsburgh Road, Butler, PA 16001, Butler, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Study Protocol: Impact of a Biophoton Therapy on Patients with Brain Disorders